CLINICAL TRIAL: NCT01125813
Title: Clinical Study to Investigate the Efficacy, Safety, and Immunogenicity of Human-cl rhFVIII in Previously Treated Patients With Severe Hemophilia A
Brief Title: Efficacy and Safety Study of Human-cl rhFVIII in PTPs With Severe Hemophilia A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GENA-08
Record Dates: First submitted 2010-05-17; First posted 2010-05-18 (Estimated); Results first posted 2013-04-22 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-08

CONDITIONS: Severe Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- human cl-rhFVIII (Experimental)
  Interventions: Biological: recombinant Factor VIII

INTERVENTIONS:
Biological: recombinant Factor VIII — intravenous infusion of factor FVIII every other day.
  Other Names: human-cl rhFVIII

SUMMARY:
This study will determine the efficacy of human-cl rhFVIII in previously treated patients with severe hemophilia A during prophylactic treatment, treatment of bleeding episodes and in surgical prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Severe hemophilia A ((FVIII:C <= 1%)
* Male subjects >= 12 years of age
* Previously treated with FVIII concentrate, at least 50 EDs
* Immunocompetent (CD4+ count > 200/ul)
* Negative for anti- HIV; if positive, viral load < 200 particles/u; or <400,000 copies/mL

Exclusion Criteria:

* Other coagulation disorder than hemophilia A
* Present of past FVIII inhibitor activity (.= 0.6 BU)
* Severe liver and kidney disease
* Receiving of scheduled to receive immuno-modulating drugs

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Oldenburg, Prof., Principal Investigator — Universitaetsklinikum Bonn
Locations (11):
- Medizinische Universitaet Wien, Vienna, Austria
- Haematological Hospital Joan Pavel, Sofia, Bulgaria
- Germany (4):
  - Werlhof Institut fuer Haemostaseologie GmbH, Hanover, Lower Saxony
  - Universitaetsklinikum, Bonn
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - SRH Kurpfalzkrankenhaus Heidelberg, Heidelberg
- United Kingdom (5):
  - Basingstoke & North Hampshire NHS Foundation Trust, Basingstoke
  - University Hospital of Wales, Cardiff
  - Royal Free Hospital, London
  - Manchester Royal Infirmary, Manchester
  - Royal Hallamshire Hospital, Sheffield

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 11 European sites beginning June 2010 and completing in January 2012.
Pre-assignment Details: 36 participants were enrolled and screened. 4 were screen failures. Therefore, 32 of the 36 enrolled were exposed to investigation product.
Groups:
- Human Cl-rhFVIII: recombinant Factor VIII : intravenous infusion of factor FVIII every other day.
Period: Overall Study
Arm/Group | Human Cl-rhFVIII
Started | 36
Completed | 30
Not Completed | 6
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Screen Failures | 4

BASELINE CHARACTERISTICS:
Arm/Group | Human Cl-rhFVIII
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 32
Region of Enrollment [Number; unit: participants]
  Austria | 1
  Bulgaria | 8
  Germany | 8
  United Kingdom | 15

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Assessment After a Total of at Least 50 EDs Per Subject at the End of the Study at 6 Months
Description: Frequency of spontaneous breakthrough bleeds/months under prophylactic treatment.
Time Frame: At least 50 Exposure Days and at least 6 months
Population: All subjects who started prophylactic treatment were evaluated.
Measure: Mean (Standard Deviation); unit: Bleeds per month
Arm/Group | Human Cl-rhFVIII
Number analyzed (Participants) | 32
Bleeds per month | 0.188 (0.307)

2. Primary Outcome: Efficacy of Treating Bleeding Episodes
Description: At the end of a bleeding episode, efficacy was assessed as:
  * Excellent: Abrupt pain relief and/or unequivocal improvement in objective signs of bleeding within approximately 8 hours after a single infusion
  * Good: Definite pain relief and/or improvement in signs of bleeding within approximately 8-12 hours after an infusion requiring up to 2 infusions for complete resolution
  * Moderate: Probable or slight beneficial effect within approximately 12 hours after the first infusion requiring more than two infusions for complete resolution
  * None: No improvement within 12 hours, or worsening of symptoms, requiring more than 2 infusions for complete resolution Efficacy was rated
Time Frame: After each bleeding episode, up to 6 month
Measure: Number; unit: Percentage of treatments
Units Other Than Participants: bleeding episodes
Arm/Group | Human Cl-rhFVIII
Number analyzed (Participants) | 32
Number analyzed (bleeding episodes) | 28
Percentage of treatments
  Excellent | 71.4
  Good | 28.6

ADVERSE EVENTS:
Arm/Group | Human Cl-rhFVIII
Serious Adverse Events (participants affected / at risk) | 2/32
Other Adverse Events (participants affected / at risk) | 3/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Human Cl-rhFVIII (N=32)
Traumatic fracture (Injury, poisoning and procedural complications) | 1
STATUS EPILEPTICUS (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Human Cl-rhFVIII (N=32)
Nasopharyngitis (Infections and infestations) | 3
Headache (Nervous system disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Pyrexia (General disorders) | 2
Contusion (Injury, poisoning and procedural complications) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less